CLINICAL TRIAL: NCT00610025
Title: Transgastric Peritoneoscopy for Evaluation of the Abdominal Wall to Direct Laparoscopic Trocar Placement
Brief Title: Minimally Invasive Trocar Placement in Obesity Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jeffrey Hazey (Other)
Collaborators: Stryker SA (Industry); Natural Orifice Surgery Consortium for Assessment and Research (Other)
Responsible Party: Sponsor-Investigator, Jeffrey Hazey, Associate Professor, Ohio State University
Organization: Ohio State University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: NOTES Trocar Study; Project 60009927; Award GRT00006515; IRB 2007H0045
Record Dates: First submitted 2007-12-26; First posted 2008-02-07 (Estimated); Last update posted 2013-02-12 (Estimated); Status verified 2013-02

CONDITIONS: Obesity
Keywords: NOTES; transgastric endoscopy; obesity surgery; Roux-en-Y surgery
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- 1 (Active Comparator): 10 patients with no previous abdominal surgeries, pre-insufflation of the abdomen using a veress needle (standard procedure for insufflating the abdomen for laparoscopic surgery)
  Interventions: Procedure: Transgastric access to the abdomen
- 2 (Active Comparator): 10 patients with history of previous abdominal surgeries, pre-insufflation of the abdomen using veress needle (standard procedure for insufflating the abdomen for laparoscopic surgery)
  Interventions: Procedure: Transgastric access to the abdomen
- 3 (Active Comparator): 10 patients with no previous history of abdominal surgeries, no veress needle pre-insufflation (insufflating the abdominal cavity through the endoscope, transgastrically)
  Interventions: Procedure: Transgastric access to the abdomen
- 4 (Active Comparator): 10 patients with history of previous abdominal surgeries, no veress needle pre-insufflation (insufflating the abdominal cavity through the endoscope, transgastrically)
  Interventions: Procedure: Transgastric access to the abdomen
- 5 (Active Comparator): 10 patients, all with no previous mid to upper abdominal surgeries, no Veress needle pre-insufflation (insufflating the abdominal cavity through the endoscope, transgastrically)
  Interventions: Procedure: Transgastric access to the abdomen
- 6 (Active Comparator): 10 patients, all with previous mid-to-upper abdominal surgeries, no Veress needle pre-insufflation, endoscopic take-down of intra-abdominal adhesions (if identified)
  Interventions: Procedure: Transgastric access to the abdomen

INTERVENTIONS:
Procedure: Transgastric access to the abdomen — Upper endoscopy, gastrotomy created with a needle knife followed by lower endoscopy.

SUMMARY:
During surgery for obesity, minimally invasive endoscopy can be performed and can assist the surgeon in determining surgical incision sites.

DETAILED DESCRIPTION:
Transgastric endoscopic access, without laparoscopic guidance, to the peritoneal cavity can be performed safely and guide trocar placement in morbidly obese patients undergoing Roux-en-y gastric bypass.

ELIGIBILITY:
Inclusion Criteria:

* Elective laparoscopic Roux-en-Y gastric bypass (LRYGB) surgery

Exclusion Criteria:

* Lack of consent
* History of previous gastric surgery
* Contraindication to upper endoscopy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2007-07; Primary Completion 2009-10 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
The achievement of safe transgastric access to the abdomen; the ability to visualize the abdominal wall to assist in safe trocar placement in the morbidly obese patient. | At surgery

SECONDARY OUTCOMES:
Bacterial contamination analysis; results compared to previous study. | Surgery

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey W Hazey, MD, Principal Investigator — The Ohio State University Medical Center/Center for Minimally Invasive Surgery
Locations (1):
- The Ohio State University Medical Center/Center for Minimally Invasive Surgery, Columbus, Ohio, United States